CLINICAL TRIAL: NCT00209521
Title: Phase 2, Randomized Study of AQUAVAN® Injection In Elective Coronary Artery Surgery With Comparison to DISOPRIVAN® Injectable Emulsion
Brief Title: Comparison of AQUAVAN® Injection to DISOPRIVAN® Injectable Emulsion for Anesthesia During Coronary Artery Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: James Vornov, MD, PhD, Guilford Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3000-0104
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Ischemic Coronary Artery Disease; Coronary Artery Bypass Surgery
Keywords: Coronary Artery Bypass Surgery; AQUAVAN® Injection; DISOPRIVAN® Injectable Emulsion.; ischemic coronary artery disease
MeSH Terms: interventions — fospropofol; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- fospropofol (Experimental)
  Interventions: Drug: fospropofol
- propofol (Active Comparator)
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: fospropofol — Using a Target Controlled Infusion (TCI) system, the target plasma concentrations of propofol to be administered from AQUAVAN were 0.7 μg/mL (sedation) and 2.5 μg/mL (maintain anesthesia).
  Other Names: fospropofol disodium; LUSEDRA; E2083; GPI-15715; AQUAVAN
  Arms: fospropofol
Drug: propofol — Using a Target Controlled Infusion (TCI) system, the target plasma concentrations of propofol to be administered from Disoprivan were 1.0 μg/mL (sedation) and 3.0 μg/mL (maintain anesthesia).
  Other Names: Disoprivan; propofol injectable emulsion
  Arms: propofol

SUMMARY:
This is an exploratory clinical trial designed to examine the efficacy, safety and tolerability of fospropofol (AQUAVAN) Injection compared to propofol (DISOPRIVAN) Injectable Emulsion when used to preoperatively sedate, induce, and maintain general anesthesia and to postoperatively sedate patients undergoing elective coronary artery surgery.

DETAILED DESCRIPTION:
This Phase 2, open-label, single-center, randomized clinical trial was designed to examine the efficacy and tolerability of AQUAVAN® Injection (hereafter, referred to as AQUAVAN) when used to preoperatively sedate, induce, and maintain general anesthesia and to postoperatively sedate patients undergoing elective coronary artery surgery. Eligible patients were randomized to either AQUAVAN or DISOPRIVAN® Injectable Emulsion (hereafter, referred to as DISOPRIVAN) following screening and prior to their arrival in the surgical suite.

On the day of surgery, after the administration a 0.5 mg/kg bolus dose of lignocaine, preoperative sedation began using the target-controlled infusion (TCI) system to target desired sedation plasma concentrations of either AQUAVAN or DISOPRIVAN, depending on the randomization schedule.

The Bispectral (BIS) Index was used to guide study drug administration; target BIS ranges were 60 to 80 for sedation and 40 to 60 for the maintenance of anesthesia. Adequate sedative/hypnotic effect during surgical anesthesia was characterized by the portion of time within the target BIS Index range versus total surgical time. Following this, during postsurgical sedation, inadequate sedative/hypnotic effect was characterized by the number, duration, and magnitude of BIS scores outside of the target range versus total postsurgical sedation time. During postsurgical sedation, the Modified Ramsey Scale was used as an additional clinical tool to evaluate the state of sedation, with an attempt to maintain the score between 3 and 5.

The overall quality of induction, maintenance and ease of control of anesthesia, and quality of sedation before and during cardiopulmonary bypass (CPB), were each graded by the anesthesiologist.

Continuous monitoring of blood pressure and heart rate were used to assess the hemodynamic effect of study drug. Hypertension and hypotension were defined as excursions of >/= 20% from the baseline value.

ELIGIBILITY:
Inclusion Criteria:

1. Patients were between the ages of 21 and 70 years, inclusive.
2. Patients were scheduled for first-time elective coronary artery bypass graft surgery, with 1 to 4 grafts planned.
3. Patients had an American Society of Anesthesiologists (ASA) Physical Classification System status of II or III.
4. Patients had a "good" left ventricular function as defined by a cardiac ejection fraction >=50% measured by cardiac catheterization or other quantitative technique.
5. Patients provided written Informed Consent after receiving a full explanation of the extent and nature of the study and were willing to comply with the study procedures.
6. Patients, if female, were surgically sterile or postmenopausal.

Exclusion Criteria:

1. Patient had prior coronary bypass grafting or other cardiac surgery.
2. Patient had uncontrolled hypertension (diastolic >110 mm Hg) or required additional intervention while hospitalized prior to surgery to control blood pressure.
3. Patient had a medical history of renal disease or creatinine >1.4 mg/dL.
4. Patient had known hemodynamically significant valvular abnormalities, except Grade 1 tricuspid or mitral insufficiency.
5. Patient had severe obesity, defined as a body mass index (BMI) >35.
6. Patient failed the Allen's Test to confirm the patency of the ulnar artery.
7. Patient had severe or uncontrolled systemic illness (e.g., pulmonary disease, cancer, endocrine abnormalities).
8. Patient had insulin-dependent diabetes.
9. Patient had a history of stroke or current neurological disease (e.g., dementia, neuropathy), as determined by the Investigator.
10. Patient had anticipated difficulties with intubation, in the judgment of the Investigator.
11. Patient had a history of alcohol abuse, as determined by the Investigator;
12. Patient had participated in an investigational drug study within 1 month prior to study start.
13. Patient had donated >300 mL of blood within 1 month prior to study start.
14. Patient had a positive medical history for drug abuse.
15. Patient had a known infection with human immunodeficiency virus (HIV), Hepatitis B, and/or Hepatitis C.
16. Patient had any history of anxiety or psychiatric illness or was currently using antidepressants, monoamine oxidase (MAO) inhibitors, anti-anxiety medications or other drugs with central nervous system (CNS) effects prior to their preoperative hospital stay.
17. Patient had uncorrected visual problems, including cataracts, glaucoma, or any significant abnormalities found on fundoscopic examination that would interfere with visual assessment of drug safety.
18. Patient had any history of adverse reaction to any opiate or anesthetic agent.
19. Patient, if male, did not agree to use an effective method of birth control between the time of screening and end of study.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2002-06; Primary Completion 2003-07 (Actual); Study Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
Median time (minutes) to loss of consciousness from induction start (reported as median and range). | Day 1

SECONDARY OUTCOMES:
Median time (minutes) to induction from start of infusion (reported as median and range). | Day 1
Time (minutes) to intubation from induction start (reported as median and range). | Day 1
Time (minutes) to extubation from end of infusion (reported as median and range). | Day 1
Time (minutes) to last suture from induction start (reported as median and range). | Day 1
Time (minutes) to full awareness from end of infusion (reported as median and range). | Day 1
Median time from End of Infusion to First Modified Ramsey Score of 3 (reported as median and range). | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: James Vornov, PhD,MD, Study Director — Eisai Inc.